CLINICAL TRIAL: NCT02596074
Title: A Phase 2, Randomized, Double-Blind, Parallel-Group Study to Assess the Pharmacodynamics, Safety/Tolerability and Efficacy of Topical Omiganan in Patients With Usual Type Vulvar Intraepithelial Neoplasia
Brief Title: Pharmacodynamics, Safety/Tolerability and Efficacy of Topical Omiganan in Patients With uVIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-010; 2015-002724-16 (EudraCT Number)
Record Dates: First submitted 2015-10-29; First posted 2015-11-04 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Usual Type Vulval Intraepithelial Neoplasia (uVIN)
MeSH Terms: interventions — Omiganan; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omiganan (CLS001) (Experimental): CLS001 topical gel, 2.5%
  Interventions: Drug: Omiganan (CLS001) topical gel
- Vehicle (Placebo Comparator): Vehicle topical gel
  Interventions: Drug: Vehicle topical gel

INTERVENTIONS:
Drug: Omiganan (CLS001) topical gel
  Arms: Omiganan (CLS001)
Drug: Vehicle topical gel
  Arms: Vehicle

SUMMARY:
To assess the pharmacodynamics, safety/tolerability and efficacy of topical Omiganan (CLS001) in patients with usual type vulvar intraepithelial neoplasia (uVIN).

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years
2. Biopsy proven uVIN, biopsies to have been taken within the last three months
3. Written informed consent to participate in the trial
4. At least one lesion that can be accurately measured (using RECIST criteria)

   * in at least one dimension with longest diameter ≥ 20mm
   * OR in two perpendicular dimensions that when multiplied together give a surface area of ≥ 120mm2 (e.g. 15mm x 8mm or 12mm x 10mm)
   * This is to ensure that 4x4mm biopsies can be performed on this lesion.

Exclusion Criteria:

1. Has any concomitant disease or significant medical conditions that would, in the opinion of the Investigator, potentially compromise the safety or compliance of the patient or may preclude the patient's successful completion of the clinical trial.
2. Clinically significant abnormalities, as judged by the Investigator, in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis) or ECG. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
3. Indication of a current active infectious disease of the vulva, other than HPV
4. Pregnant, breast feeding or trying to conceive
5. Active treatment for uVIN (i.e. surgical excision, lasertherapy, imiquimod, photodynamic therapy) within the previous month
6. Patients receiving immunosuppressive therapy
7. HIV positive or transplant patients
8. Any condition that in the opinion of the investigator could interfere with the conduct of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2017-03-07 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics (HPV Viral Load Assessment) | 24 Weeks
  Assessment of target lesions by quantitative PCR including HPV genotyping in swabs and biopsies
Pharmacodynamics (Local Immunity Status) | 24 Weeks
  Histological changes in immune cells in the mucosa/submucosa
Clinical Assessment (Lesions by RECIST) | 24 Weeks
  Efficacy assessment of lesions by RECIST
Clinical Assessment (Percent clearance of Lesions) | 24 Weeks
  Efficacy assessment of percent clearance of lesions
Clinical Assessment (Sum of the longest diameter (SLD)) | 24 Weeks
  Efficacy assessment of the sum of the longest diameter (SLD))
Clinical Assessment (Histology) | 24 Weeks
  Efficacy assessment of the histology (regression of uVIN to no dysplasia)

SECONDARY OUTCOMES:
Safety and Tolerability (Adverse Events) | 48 Weeks
  Adverse Events will be collected throughout the study
Safety and Tolerability (Laboratory Safety Testing) | 48 Weeks
  Laboratory Samples will be collected throughout the study
Safety and Tolerability (12-Lead ECGs) | 48 Weeks
  12-Lead ECGs will be performed throughout the study
Safety and Tolerability (Vital Signs) | 48 Weeks
  Vital Signs will be collected throughout the study
Pharmacokinetics (Area Under the Curve) | 12 Weeks
  AUC will be computed
Pharmacokinetics (Maximum Plasma Concentration) | 12 Weeks
  Cmax will be determined
Pharmacokinetics (Tmax) | 12 Weeks
  Tmax will be determined

CONTACTS AND LOCATIONS:
Overall Officials: J. (Koos) Burggraaf, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- LUMC/Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Rijsbergen M, Rijneveld R, Todd M, Feiss GL, Kouwenhoven STP, Quint KD, van Alewijk DCJG, de Koning MNC, Klaassen ES, Burggraaf J, Rissmann R, van Poelgeest MIE. Results of phase 2 trials exploring the safety and efficacy of omiganan in patients with human papillomavirus-induced genital lesions. Br J Clin Pharmacol. 2020 Nov;86(11):2133-2143. doi: 10.1111/bcp.14181. Epub 2020 Sep 28. PMID 31755993